CLINICAL TRIAL: NCT01898377
Title: Open-label, Multicenter Phase II Study of Combination Therapy of Imatinib Mesylate and Mycophenolate Mofetil in Children With Steroid-Refractory Sclerotic/Fibrotic Type Chronic Graft-versus-host Disease
Brief Title: Imatinib Mesylate and Mycophenolate Mofetil for Steroid-Refractory Sclerotic/Fibrotic cGVHD in Children
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: New treatment option introduced for patients with the study indication
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUCH-1301
Record Dates: First submitted 2013-06-05; First posted 2013-07-12 (Estimated); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Chronic Graft-versus-host Disease
Keywords: Children; Chronic graft-versus-host disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Imatinib Mesylate; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imatinib mesylate, Mycophenolate mofetil (Experimental): MMF 15-20mg/kg (Max 1 g) bid + Imatinib mesylate qd
  * Dose of imatinib : starting dose 260 mg/m2/d (Max. 400 mg)
  * Imatinib dose adjustment : Dose is adjusted according to the guidelines if there is serious adverse event, toxicity, or intolerance.
  Interventions: Drug: Imatinib mesylate, Mycophenolate mofetil

INTERVENTIONS:
Drug: Imatinib mesylate, Mycophenolate mofetil
  Other Names: Glivec, Cellcept

SUMMARY:
In this study we will combine mycophenolate mofetil and imatinib mesylate to treat steroid-refractory sclerotic/fibrotic type chronic graft-versus-host disease (GVHD) to see the response rate and to find the safety of combination.

DETAILED DESCRIPTION:
Sclerotic/fibrotic type chronic GVHD is one of the most severe forms of the disease and is frequently refractory to standard treatment approaches. Imatinib mesylate, a tyrosine kinase inhibitor, has been shown to be effective in patients with sclerotic/fibrotic type chronic GVHD by strongly inhibiting both PDGF (Platelet-derived growth factor) and TGF-β (transforming growth factor-β) intracellular signaling, which is responsible for the expression of extracellular matrix genes.

Mycophenolate mofetil (MMF) is one of effective agent for the treatment of chronic graft-versus-host disease. MMF is rapidly absorbed after oral administration and hydrolyzed to the active metabolite, MPA (mycophenolic acid). MPA selectively inhibits inosine monophosphate dehydrogenase, blocking the pathway of purine synthesis in T and B lymphocytes. In this study we will combine MMF and imatinib mesylate to treat steroid-refractory sclerotic/fibrotic type chronic GVHD to see the response rate and to find the safety of combination.

ELIGIBILITY:
Inclusion criteria

* Patients must have a diagnosis of chronic GVHD with fibrotic/scleroderma-like features. This diagnosis can be made clinically or by histopathology.
* Patients must have active disease with at least one of the following manifestations: skin sclerosis, symptomatic bronchiolitis obliterans, extensive lung fibrosis, pathologically demonstrated visceral fibrotic involvement of the gut.
* Patients with corticosteroid refractory or dependant cGVHD are eligible. Steroid-refractory chronic GVHD is defined as chronic GVHD of sustained severity during the last full month during which the patients received the equivalent of prednisone 0.5 mg/kg or more per day or 1 mg/kg or more every other day.
* Age under 21 years old

Exclusion criteria

* Patients who have had chemotherapy, radiotherapy within 4 weeks prior to entering the study.
* Patients who have not recovered from adverse events.
* Prior treatment with imatinib mesylate or other tyrosine kinase inhibitor after the date of transplant.
* Patients on pregnancy or lactating

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2013-08; Primary Completion 2018-02-14 (Actual); Study Completion 2018-02-14 (Actual)

PRIMARY OUTCOMES:
Overall (complete and partial) response rate | 1 year
  Response evaluation will be performed every 3 months during the treatment by comprehensive response criteria based on NIH criteria. The complete and partial response categories apply only to organs that have measurable and reversible GVHD-related abnormalities at baseline.
  * Complete response (CR): Resolution of all signs and symptoms of chronic GVHD
  * Partial response (PR) : Improvement (at least 1 clinical score reduction, see Appendix 2) in 1 or more organs of involvement and no evidence of worsening in any organ
  * Objective response (OR): Either CR or PR

SECONDARY OUTCOMES:
Evaluate the safety profile of MMF plus imatinib mesylate | 1 year
  All adverse events will be recorded on the "Adverse Events CRF" with the following information
  * Severity grade (NCI CTCAE ver. 4.0)
  * Relationship to the study drug
  * Duration (start and end dates or if continuing at final exam)
  * Whether it constitutes a serious adverse event (SAE)
Evaluate the quality of life (QOL) | 1 year
  The assessment of QOL will be performed at baseline and every 3 months till 1 year with Lee cGVHD Symptom Scale.
Discontinuation of steroid | 1 year
  * Based on the response during study period, investigators could modify the dosage of concomitant immunosuppressive agents in the same manner as corticosteroid.
  * The rate of discontinuation among patients and the dose change from baseline of each patient.
Overall survival rate | 1 year
  For survival outcome, Kaplan-Meier method will be used for estimation.

CONTACTS AND LOCATIONS:
Overall Officials: Hyoung Jin Kang, MD, Ph.D, Principal Investigator — Seoul National University Children's Hospital
Locations (1):
- Seoul National University Children's Hospital, Seoul, Chongno-gu, South Korea